CLINICAL TRIAL: NCT03483467
Title: Pilot Study - Effectiveness of Omnigen in Addition to Standard Treatment in Treating Diabetic Foot Ulcers (DFU)
Brief Title: Omnigen DFU Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Collaborators: NuVision Biotherapies Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DHRD/2017/042
Record Dates: First submitted 2018-03-16; First posted 2018-03-30 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): Application of Omnigen
  Interventions: Other: Omnigen
- 2 (Placebo Comparator): Dummy Omnigen Packaging
  Interventions: Other: Dummy Packaging

INTERVENTIONS:
Other: Omnigen — For those randomised onto the investigational arm, a dual layer of the Omnigen product will be applied at baseline and at every fortnightly trial visit until healing or the end of the 12 week period whichever occurs first, according to the standard study procedure.
  Arms: 1
Other: Dummy Packaging — For those randomised into the control arm, dummy packaging will be opened at the time of application of standard of care, to ensure the same experience is received to those on the experiential arm.
  Arms: 2

SUMMARY:
The Omnigen Pilot study aims to provide an evidence base for Omnigen as a treatment for Diabetic Foot Ulcers (DFU). It aims to achieve this by tailoring a regenerative therapy used for ocular surface repair to provide proactive non-surgical wound management of Diabetic Foot Ulcers (DFU).

DETAILED DESCRIPTION:
This pilot study is designed as a multi-centre prospective, patient and observer blind, randomised controlled trial, recruiting patients from two clinical centres across the East Midlands; Derby Teaching Hospitals NHS Foundation Trust (DHFT) and Nottingham University Hospitals NHS Trust (NUH).

Eligible patients will be approached within diabetic foot clinics by their usual clinical carers to determine whether they are interested in participating in the study. They will be provided with written information about the study and the researcher will explain the study verbally to them and address any questions and concerns the patient may have. Patents will be given at least 24 hours to consider taking part in the trial before signing a consent form.

After informed consent has been given, baseline information will be collected. This will include demographic information, medical history and concomitant medication. eGFR and HbA1c will also be collected if not done within previous 3 months as part of standard care. The baseline wound status, assessment of ulcer infection according to Infectious Diseases Society of America (IDSA) criteria, peripheral pulses, neuropathy and ankle brachial pressure index will also be taken.

Participants will then be randomised to receive either standard of care or Omnigen graft with standard of care. Staff administering the Omnigen product will be aware of which treatment the participant is receiving however the participant and the research staff conducting the healing assessments will be blinded to their treatment allocation. Therefore the participant and the assessors will be blinded to the treatment given in order to minimize any bias in the collection of healing outcome data. For those randomized into the control arm, 'Dummy Packaging' will be used to ensure the blind is maintained.

Patients will be seen two weekly from their baseline visit until healing for up to 12 weeks and at 2 weeks post healing in those that heal. If a participant's foot ulcer heals before the final 12 weeks visit, they will attend a healing confirmation visit two weeks post the original heal date, however will not be required to attend any further fortnightly visits until the final blinded assessment visit at week 12 . If the participant's foot ulcer has not healed at 12 weeks then a blinded assessment should still be conducted at this time point.

Data is collected using the Dacima Clinical Suite Electronic Data Capture (EDC) software (Dacima Software Inc.)

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes (according to WHO criteria) aged 18 years or over
* At least one full thickness ulcer below the malleolus of either foot, present for 4 weeks or more.
* At least one palpable pulse on the foot of the index limb or an ABPI >0.9
* Minimum ulcer diameter of 5 mm
* Maximum ulcer diameter of 20 mm.
* Able to attend clinic on a fortnightly basis

Exclusion Criteria:

* eGFR <20
* HbA1c >108
* Planned revascularisation during the course of the study or within the 4 weeks preceding the start of the study
* An ulcer of aetiology other than diabetes
* Depth of ulcer to bone, suspected or confirmed osteomyelitis
* Severe infection of the index ulcer
* Active Charcot of the foot of the index ulcer
* The need for negative pressure wound therapy
* On treatment with systemic steroids at a dose > equivalent of 5mg prednisolone for more than 5 days and/or systemic cytotoxic agents
* Unwilling or unable to attend all trial visits.
* Unwilling or unable to give written informed consent.
* Lacks the mental capacity to give consent
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, may influence the result of the trial or the participant's ability to participate in the trial
* Participants who have participated in another research trial involving a wound healing product within the past 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-03-11 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-06-27 (Actual)

PRIMARY OUTCOMES:
The primary outcome is wound healing (defined as full epithelialisation without drainage maintained for 2 weeks) within 12 weeks of starting study treatment. | 12 weeks
  To assess the whether higher proportion of wounds heal at 12 weeks in the investigational arm to the control arm - assessed by confirmation of healing at 12 week visit.

SECONDARY OUTCOMES:
Overall reduction in wound size (surface area, assessed by acetate tracing) | 12 weeks
  To assess the whether higher proportion of wounds reduce in size at 12 weeks in the investigational arm to the control arm - assessed by comparing acetate tracing in each arm.
Time to healing (weeks) for those that heal within 12 weeks, | 12 weeks
  To assess the whether higher proportion of wounds heal at 12 weeks in the investigational arm to the control arm - assessed by proportion of confirmation of heeling visits conducted at 12 weeks within each arm.
Proportion of wounds healed within 6 weeks | 6 weeks
  To assess the whether higher proportion of wounds heal at 6 weeks in the investigational arm to the control arm - assessed by proportion of confirmation of heeling visits conducted at 6 weeks within each arm.
Adverse events (safety) including major and minor amputations and hospitalisation | 12 weeks
  To assess the safety of the intervention of Omnigen in comparison to standard of care. Review of SAEARs.
Incidence of secondary infection | 12 weeks
  To assess the safety of the intervention of Omnigen in comparison to standard of care. Review of SAEARs.
Feasibility of recruitment | 12 weeks
  To assess the feasibility of the study in regards to recruitment for a future full RCT. Recruitment rate, reasons for patients not randomising and reasons for investigators not randomising. Screening logs/protocol deviations.
Pain in the area of the ulcer as assessed by patient completed VAS | 12 weeks
  To assess pain of ulcer through completion of VAS at every fortnightly visit to identify if pain reduces at a higher rate on the interventional arm than the control arm.
Effectiveness of participant blind | 12 weeks
  To assess whether the blinding to arm allocation has been successful with the use of dummy packaging or whether the participants are able to identify which treatment they have received. This will be done by completion of a participant questionnaire at the end of the study.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University Hospitals Derby and Burton, Royal Derby Hospital, Derby
  - University of Nottingham Teachig Hospitals, City Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: No